CLINICAL TRIAL: NCT05425186
Title: Analysis of Reliability and Validity of Urdu Version of Rivermead Extended Activities of Daily Life Among Pakistani Population
Brief Title: A Reliability and Validity Study: Urdu Version of Rivermead Extended Activities of Daily Life
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Other Study IDs: REC-FSD-00263
Record Dates: First submitted 2022-06-15; First posted 2022-06-21 (Actual); Last update posted 2022-06-21 (Actual); Status verified 2022-06

CONDITIONS: Neurological Disorder
Keywords: Rivermead Extended Activities of Daily Life; Urdu Version; Reliability; Validity; Neurological Disorder
MeSH Terms: conditions — Nervous System Diseases

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The goal of this study is to translate and culturally adapt Rivermead Extended Activities of Daily Life into the Urdu language and to evaluate its reliability and validity in the Pakistani neurological rehabilitation population. Also assess its correlation with Memory and Concentration Test, The Barthel Index, and The index of French activities.

DETAILED DESCRIPTION:
As per the preceding commendation, Rivermead Extended Activities of Daily Life will be deciphered into the Urdu dialect from its English adaptation and adjusted socially in Pakistan. Among the neurological rehabilitation population, Rivermead Extended Activities of Daily Life will be distributed in 100 patients enrolled by comfort inspecting strategy beneath the pre-defined incorporation and avoidance criteria after marking assent shapes. For testing inter-observer unwavering quality and intra-observer unwavering quality of Rivermead Extended Activities of Daily Life, Memory and Concentration Test, index of French activities, and Barthel Index surveys will be managed by spectator, on the same day, with a time interval of 2 hours between 1st and 2nd readings. As for the 3rd readings, it will be carried out after seven days by the first observer, for intra-observer appraisal. Statistical Package of Social Sciences computer program has been utilized for information passage and examination. Inner consistency will be analyzed with Cronbach alpha esteem. Test-retest unwavering quality will be surveyed by utilizing an intra-class relationship coefficient. The Rivermead Extended Activities of Daily Life will be assessed for content validity, construct validity, criterion validity, and responsiveness.

ELIGIBILITY:
Inclusion Criteria:

* Patients from Rehabilitation centers mainly outpatients; with more or severe impairments due to neurological /neuro-muscular diseases.
* Patient should be in a stable state unlikely to change over 2- weeks.
* Patient should score 18/28 short orientation-memory-concentration test; indicating a reasonable cognitive and communicative ability.

Exclusion Criteria:

* People not suffering from any neurological impairment.
* Scorning less than 18/28 on short orientation-memory-concentration test.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: We targeted the Pakistani stroke and head injury population received rehabilitation for neurological impairments in our study.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2021-05-30 (Actual); Primary Completion 2022-07-10 (Estimated); Study Completion 2022-07-12 (Estimated)

PRIMARY OUTCOMES:
Rivermead Extended Activities of Daily Life | 1st day
  Rivermead Extended Activities of Daily Life having 10 things in it is in fact could be a complete independent community survival scale, covering all the fundamental independent living fashion needs. Restoration administrations are pointed at accomplishing social autonomy within the community, on the off chance that conceivable, and must utilize an fitting degree of Rivermead Extended Activities of Daily Life when they are assessed themselves.
Memory and Concentration Test | 1st day
  The Brief Introduction Memory and Concentration Test is one of numerous tests of memory and concentration. It has the advantage of having decently culture-free substance. In expansion, it covers moderately restricted zones of cognition: is the individual arranged; can the individual center on a brief errand; and can the person learn and keep in mind a number of basic things.
Frenchay Activities Index | 1st day
  The Frenchay Activities Index is a measure of instrumental activities of daily living for use with patients recovering from stroke.
Barthel Index | 1st day
  The Barthel index is used to assess disability and to monitor changes in disability over time. The scoring method takes into account whether the person evaluated receives help while doing each task.

CONTACTS AND LOCATIONS:
Overall Officials: Muhammad Kashif, Study Chair — Riphah International University
Locations (1):
- Ripah International University, Faisalabad, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No